CLINICAL TRIAL: NCT01295177
Title: Topic Insulin Accelerates Wound in Diabetes
Brief Title: Topic Insulin Accelerates Wound Healing in Diabetes
Acronym: insulin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: mhmelolima@gmail.com, unicamp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INSULIN22
Record Dates: First submitted 2011-02-03; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus; Wounds
Keywords: wound healing; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vehicle cream (Placebo Comparator): Intervention: Placebo cream vehicle. Patients with wounds for more than 3 months without infection. These patients were treated with placebo cream (cream with the same constitution but without insulin). The placebo cream vehicle was used for 8 weeks.
  Interventions: Drug: topic cream insulin
- cream insulin (Placebo Comparator): Intervention: insulin cream. Patients with wounds for more than 3 months without infection. These patients were treated with insulin cream (cream with the same constitution but with insulin). The insulin cream was used for 8 weeks.
  Interventions: Drug: topic cream insulin

INTERVENTIONS:
Drug: topic cream insulin — Intervention: Placebo cream versus insulin cream. Patients with wounds for more than 3 months without infection. These patients were treated with placebo cream or insulin cream. The placebo or insulin were used for 8 weeks.
  Other Names: wound healing; insulin cream; diabetes

SUMMARY:
The purpose of this study is to determine whether topic insulin is effective to accelerates wound healing in diabetes patients

DETAILED DESCRIPTION:
Wound healing is impaired in diabetes mellitus, but the mechanisms involved are not well established. The purpose of this study was to investigate the effect of a topic insulin cream on wound healing in diabetic patients. age eligible for study:18 years old-older gender eligible for study:both accepts healthy volunteers:no have a proband with T1DM or T2DM. A proband is an individual with more than one year of diagnosis.

have proband with a wound that is difficult to be healed for at least three months.

patients with serum creatinine <1.5mg/dl Does not satisfy the above inclusion criteria infection diagnosed wound patients with cellulitis, venous stasis, inadequate perfusion, osteomyelitis and patient's inability to attend clinics for follow up

ELIGIBILITY:
Inclusion Criteria:

age eligible for study:18 years old-older gender eligible for study:both accepts healthy volunteers:no have a proband with T1DM or T2DM. A proband is an individual with more than one year of diagnosis. have proband with a wound that is difficult to be healed for at least three months.

patients with serum creatinine <1.5mg/dl

Exclusion Criteria:

Does not satisfy the above inclusion criteria infection diagnosed wound patients with cellulitis, venous stasis, inadequate perfusion, osteomyelitis and patient's inability to attend clinics for follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
% of Wound healing closing measured each week | 7 days

SECONDARY OUTCOMES:
Complete wound healing | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena M Lima, PhD, Study Chair — University of Campinas (UNICAMP); Mario J Saad, MD PhD, Principal Investigator — University of Campinas (UNICAMP)

REFERENCES:
- [Derived] Lima MH, Caricilli AM, de Abreu LL, Araujo EP, Pelegrinelli FF, Thirone AC, Tsukumo DM, Pessoa AF, dos Santos MF, de Moraes MA, Carvalheira JB, Velloso LA, Saad MJ. Topical insulin accelerates wound healing in diabetes by enhancing the AKT and ERK pathways: a double-blind placebo-controlled clinical trial. PLoS One. 2012;7(5):e36974. doi: 10.1371/journal.pone.0036974. Epub 2012 May 25. PMID 22662132